CLINICAL TRIAL: NCT03292731
Title: Relationship Between Plasma Concentration of (Hydroxyprogesterone Caproate) 17-OHPC and Preterm Birth
Brief Title: Relationship Between Plasma Concentration of Hydroxyprogesterone Caproate (17-OHPC) and Preterm Birth
Acronym: PRO
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: grant funding cycle ended
Sponsor: Steve N. Caritis, MD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Steve N. Caritis, MD, Professor, Department of OB/Gyn/RS, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO16110007; U54HD047905-11 (NIH); STUDY19020368 (Other: PittPRO)
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Safety

STUDY DESIGN:
Intervention Model Description: An open labelled rct for secondary analysis of safety of 500 mg dose. A pharmacodynamic study of 17-OHPC concentration and rate of sPTB
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- hydroxyprogesterone caproate 500 mg (Experimental): For safety assessment of the 500 mg dose, subjects will be randomized to the 500 mg dose of 17-OHPC.
  Interventions: Drug: Safety study of 500 mg dose.
- hydroxyprogesterone caproate 250 mg (Active Comparator): For safety assessment of the 500 mg dose, subjects will be randomized to the 250mg dose of 17-OHPC.
  Interventions: Drug: 17-Hydroxyprogesterone caproate 250mg or 500 mg.
- Ancillary cohort 250 mg dose (Active Comparator): Receiving 250 mg as part of routine care
  Interventions: Drug: 17-Hydroxyprogesterone caproate 250mg or 500 mg.

INTERVENTIONS:
Drug: 17-Hydroxyprogesterone caproate 250mg or 500 mg. — For the pharmacodynamic study, subjects receiving either 250mg or 500 mg dose will be studied to relate the plasma concentration at 26-30 to the rate of sPTB. For the safety study, subjects will be randomized to either the 250mg or 500 mg dose.
  Other Names: pharmacodynamic
  Arms: Ancillary cohort 250 mg dose; hydroxyprogesterone caproate 250 mg
Drug: Safety study of 500 mg dose. — Subjects randomized to 250 mg or 500 mg dose
  Other Names: safety
  Arms: hydroxyprogesterone caproate 500 mg

SUMMARY:
The study plans to determine the relationship between plasma concentrations of 17-OHPC hydroxyprogesterone caproate (17-OHPC) and the rate of preterm birth. The study is an open label study of pregnant women with one or more prior spontaneous preterm births who are receiving either 250mg of 500 mg of 17-OHPC as a weekly single injection. The safety of the 500 mg dose will also be assessed.

DETAILED DESCRIPTION:
The study will determine the association between plasma concentrations of 17-OHPC (hydroxyprogesterone caproate) and the rate of preterm birth and will evaluate the impact of several potential covariates on plasma concentrations of 17-OHPC and its efficacy. 17-OHPC (hydroxyprogesterone caproate) administration has proven effective in reducing preterm births in high risk groups but the current dose of 250mg administered intramuscular (IM ) is thought to be an inadequate for a substantial portion of women receiving the therapy. The potential benefit of identifying a therapeutic concentration range and of optimizing the dosage of 17-OHPC are substantial.

One cohort of pregnant subjects with a history of a prior spontaneous preterm birth with be randomized to either the 250mg or 500mg weekly intramuscular injections. All subjects will have trough blood samples collected immediately prior to their second injection of the 17-OHPC, at 26-30 weeks (but only after a minimum of 7 injections have been administered) , 6-9 weeks later and at the time of delivery. Another tube of maternal blood will be collected during one of the scheduled blood samples for genotyping. A cord blood specimen will also be collected and with consent, a cord blood specimen will be collected for genetic studies of the infant. Investigators will also collect a small sample of the placenta after delivery.

In order to enhance sample size for this trial, investigators will also enroll a second cohort of subjects (ancillary cohort) who are not in the randomized clinical trial (RCT) described above. Women already receiving 250 mg 17-OHPC weekly from their healthcare provider as part of their standard of care will be approached prior to 26 weeks gestation. This will be an observational cohort and subjects enrolled in the ancillary cohort will not be randomized, as they are already receiving the 250 mg dose. Research staff will not administer the study drug to subjects enrolled in the ancillary cohort. These subjects will be asked to provide two blood samples: one at 26-30 weeks and one 6-9 weeks later, which will be utilized to address the primary objective of the study.

In response to the addition of the ancillary cohort, randomization for subjects in the RCT will be 2:1 for the 500 mg vs the 250 mg dose. The ancillary study will be implemented initially at the UPITT site only but may be expanded to other sites, as required.

ELIGIBILITY:
1. Randomized Clinical Trial Eligibility Criteria:

   Inclusion Criteria:
   * pregnant with a prior preterm birth 16 0/7-35 6/7 weeks from spontaneous labor or preterm premature rupture of membranes(PPROM),
   * current gestational age <22 weeks,
   * pregnant with one baby
   * age between 18-45 years
   * able to give consent and undergo study procedures

   Exclusion Criteria:
   * plans for cerclage at enrollment, plan for progesterone treatment other than study medications at enrollment
   * known fetal anomaly or chromosomal anomaly that could affect gestational age at delivery
   * malformation of the uterus or known cervical length <2.5cm
   * participation in another trial that may affect gestational age at delivery
   * planned delivery where outcome data cannot be collected
   * medical or obstetrical complication that may affect gestational age at delivery, such as active ulcerative colitis, liver tumors, liver disease/failure, renal disease/failure, undiagnosed vaginal bleeding unrelated to pregnancy, or hypertension requiring 2 or more agents
   * Current or history of thrombosis or thromboembolic disorders
   * known or suspected breast cancer, other hormone-sensitive cancer, or a history of these conditions
   * moderately severe depression (PHQ-9 score ≥ 15, EPDS score of >13, or suicidal ideation)
2. Ancillary Cohort Eligibility Criteria:

Inclusion Criteria:

* Pregnant female with documented prior birth between 16 0/7- 35 6/7 week gestation from spontaneous preterm labor or preterm premature rupture of membranes
* Receiving 250 mg 17-OHPC weekly- must be compliant with that treatment based on interview and reviewing the medical record
* Gestational age (GA) <26 weeks, based on study determined GA
* Singleton gestation
* Age between 18 - 45 years
* Able to give informed consent and undergo study procedures

Exclusion Criteria:

* Inclusion in the RCT of 250 vs 500 mg OPRC study
* Cerclage in place
* Plan for progesterone treatment other than study medication
* Known major fetal anomaly or chromosomal anomalies that might affect gestational age at delivery
* Malformation of uterus (uterine didelphus, septate uterus or bicornuate uterus) or known cervical length <2.5 cm
* Participation in another trial that may affect gestational age at delivery
* Planned delivery at other institution where pregnancy outcome data cannot be obtained
* Medical or obstetrical complication that might affect gestational age at delivery, such as active ulcerative colitis, liver tumors, liver disease/failure, renal disease/failure, undiagnosed vaginal bleeding unrelated to pregnancy, or hypertension requiring 2 or more agents
* Current or history of thrombosis or thromboembolic disorder.
* Known or suspected breast cancer, other hormone-sensitive cancer, or a history of these conditions.
* Moderately severe depression (PHQ-9 score ≥15, EPDS score of >13, or suicidal ideation)- based on criteria in the RCT

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Study of pregnant participants
Enrollment: 159 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve N Caritis, MD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - University of Pittsburgh-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data to be shared include plasma 17-OHPC concentrations , rates of sPTB, and data on maternal adverse effects and neonatal outcomes
Supporting Information: Study Protocol
Time Frame: These data will be eligible to the recruiting centers after the main data are published. they will have 18 months to request secondary analyses . other researchers will have access to the data after that period.
Access Criteria: To be determined by the OPRC steering committee.

REFERENCES:
- [Derived] Caritis SN, Costantine MM, Clark S, Stika CS, Kiley JW, Metz TD, Chauhan SP, Venkataramanan R; Eunice Kennedy Shriver National Institute of Child Health and Human Development Obstetric-Fetal Pharmacology Research Centers Network. Relationship between plasma concentration of 17-hydroxyprogesterone caproate and gestational age at preterm delivery. Am J Obstet Gynecol MFM. 2023 Jul;5(7):100980. doi: 10.1016/j.ajogmf.2023.100980. Epub 2023 Apr 24. PMID 37100349

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydroxyprogesterone Caproate 250 mg RCT Component: Pregnant subject will be randomized either to 250mg or 500 mg of hydroxyprogesterone caproate Intramuscular .
- Hydroxyprogesterone Caproate 500 mg RCT Component: Participants wil be randomized to either 250 mg or a 500 mg dose
- 250 mg 17-OHPC Ancillary Component: subjects already on 17-OHPC will be enrolled and followed
Period: Overall Study
Arm/Group | Hydroxyprogesterone Caproate 250 mg RCT Component | Hydroxyprogesterone Caproate 500 mg RCT Component | 250 mg 17-OHPC Ancillary Component
Started | 67 | 76 | 16
Completed | 63 | 65 | 15
Not Completed | 4 | 11 | 1
Not completed — Protocol Violation | 4 | 11 | 1

BASELINE CHARACTERISTICS:
Population: Includes those who were compliant with study procedures and continued treatment
Groups:
- Hydroxyprogesterone Caproate 250 mg RCT Cohort: Pregnant subjects randomized to 250mg of hydroxyprogesterone caproate RCT cohort
- Hydroxyprogesterone Caproate 500 mg RCT Cohort: Pregnant subjects randomized to 500 mg of hydroxyprogesterone caproate RCT cohort
- Hydroxyprogesterone Caproate 250 mg Ancillary Cohort: Pregnant subjects receiving 250 mg of hydroxyprogesterone caproate Ancillary cohort
- Total: Total of all reporting groups
Arm/Group | Hydroxyprogesterone Caproate 250 mg RCT Cohort | Hydroxyprogesterone Caproate 500 mg RCT Cohort | Hydroxyprogesterone Caproate 250 mg Ancillary Cohort | Total
Number analyzed (Participants) | 67 | 76 | 16 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 67 | 76 | 16 | 159
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — age in years stated by participant
  years | 30.8 (5.5) | 30.5 (5.4) | 32.7 (3.3) | 30.8 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 76 | 16 | 159
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 13 | 0 | 20
  White | 56 | 61 | 16 | 133
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67 | 76 | 16 | 159

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between 17-OHPC Concentration and Spontaneous Preterm Birth - A Concentration-Response Analysis
Description: relationship between the rate of spontaneous preterm birth ( delivery < 37 weeks) and drug concentration obtained at 26-30 weeks among those with a blood sample and adherent to study protocol (n=116)
Time Frame: 26-30 week blood sample after a minimum of 7 injections among those with a blood sample and compliant with protocol(n=116)
Population: the primary outcome was pre-specified as only applying to those receiving either 250 mg or 500 mg dose and having a blood sample drawn according to protocol and having received at least 7 injections (n=116). The number of sPTBs is listed by group in the outcome table.
Measure: Count of Participants; unit: Participants
Groups:
- Ancillary -250 mg: Ancillary group receiving 250 mg not randomized
- RCT Group 250 mg Dose: this group was randomized to 250 mg dose
- RCT Group -500 mg Dose: This group randomized to 500 mg
- Summarized OHPC: Includes all 17-OHPC values across groups
Arm/Group | Ancillary -250 mg | RCT Group 250 mg Dose | RCT Group -500 mg Dose | Summarized OHPC
Number analyzed (Participants) | 14 | 48 | 54 | 116
Participants | 1 | 9 | 12 | 22
Statistical Analysis 1: Comparison: Ancillary -250 mg vs RCT Group 250 mg Dose vs RCT Group -500 mg Dose vs Summarized OHPC; logistic regression comparing drug concentration to the rate of sPTB; Test type: Other; p = 0.96, Regression, Logistic — adjusted for cerclage; adjusted for cerclage; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.93 to 1.08]

2. Primary Outcome: Survival A
Description: days from first injection to spontaneous preterm delivery
Time Frame: time in days from first injection to spontaneous preterm delivery
Population: Subjects with a blood sample and no more than two missed injections
Measure: Mean (Standard Deviation); unit: days
Groups:
- Ancillary-250 mg: ancillary group received 250 mg dose
- RCT Group 250 mg Dose: thiw group was randomized to 250 mg
- Summarized OHPC: includes all 17-OHP{C values across groups
Arm/Group | Ancillary-250 mg | RCT Group 250 mg Dose | RCT Group -500 mg Dose | Summarized OHPC
Number analyzed (Participants) | 14 | 48 | 54 | 116
days | 150 (37) | 144 (17) | 145 (19) | 145 (21)
Statistical Analysis 1: Comparison: Ancillary-250 mg; Test type: Other; p = 0.05, Regression, Linear; Slope = 1.11, 95% CI 2-sided [0.00 to 2.23]

3. Primary Outcome: Survival B
Description: days from when the 26-30 week blood sample was obtained to the gestation at spontaneous preterm birth. All blood samples were obtained after at least 7 injections were give by which time steady state would have been achieved. This analysis was limited to those with a 26-30 week blood sample who were compliant with the protocol
Time Frame: days from blood sample time to spontaneous preterm delivery
Population: This analysis was limited to those 116 subjects with a 26-30 week blood sample who were compliant with the protocol regardless of group
Measure: Mean (Standard Deviation); unit: days
Groups:
- Ancillary -250 mg: days from blood draw to preterm birth
- RCT Group 250 mg Dose: group randomized to 250 mg
- RCT Group -500mg Dose: group randomized to 500 mg
Arm/Group | Ancillary -250 mg | RCT Group 250 mg Dose | RCT Group -500mg Dose | Summarized OHPC
Number analyzed (Participants) | 14 | 48 | 54 | 116
days | 74 (15) | 73 (18) | 73 (19) | 73 (18)
Statistical Analysis 1: Comparison: Summarized OHPC; Test type: Other; p = 0.022, Regression, Linear; Slope = 1.56, 95% CI 2-sided [0.25 to 2.87]

4. Secondary Outcome: Composite Neonatal Outcome
Description: Composite NN outcome (fetal death, neonatal death (NND), respiratory distress syndrome, bronchopulmonary dysplasia, necrotizing enterocolitis, intraventricular hemorrhage 3 or 4, retinopathy of prematurity, hypoxic-ischemic encephalopathy, seizures.) and NICU admission
Time Frame: till discharge from nicu up to 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Ancillary- 250 mg Dose: group received 250 mg dose not randomized
- RCT - 250 mg Dose: Group randomized to 250 mg dose
- RCT - 500 mg Dose: Group randomized to 500 mg dose
- Summarized 17-OHPC: Includes data across all groups
Arm/Group | Ancillary- 250 mg Dose | RCT - 250 mg Dose | RCT - 500 mg Dose | Summarized 17-OHPC
Number analyzed (Participants) | 15 | 65 | 66 | 146
Participants | 3 | 10 | 12 | 25
Statistical Analysis 1: Comparison: RCT - 250 mg Dose vs RCT - 500 mg Dose; Only RCT subjects utilized in neonatal safety analysis; Test type: Superiority; p = 0.82, Fisher Exact — no adjustments

5. Secondary Outcome: NICU Admission
Description: Infants admitted to the NICU
Time Frame: any admission to the NICU from time of delivery to time of discharge from the hospital up to 30 days or transfer to another facility
Population: Only includes those neonates exposed to 17-OHPC who's mothers were randomized to either the 250 mg or 500 mg dose . Those in the ancillary study were excluded from this analysis
Measure: Count of Participants; unit: Participants
Groups:
- 250 mg Dose: safety of 250 mg dose
- 500 mg Dose: safety of 500mg dose
- All RCT Groups: Includes all subjects in the RCT
Arm/Group | 250 mg Dose | 500 mg Dose | All RCT Groups
Number analyzed (Participants) | 65 | 66 | 131
Participants | 11 | 16 | 27

6. Secondary Outcome: Comparison of Plasma Concentration of 17-OHPC According to Dose
Description: Plasma concentrations of 17-OHPC after 250 or 500 mg dose. Subjects were compliant with protocol up to the 26-30 week blood draw and had a blood sample available . This included subjects with indicated preterm birth and was not limited to those with spontaneous PTB. Plasma concentration among those receiving the 250 mg dose are compared to those receiving 500 mg dose.
  Those receiving the 250 mg dose include both the RCT and ancillary groups.
Time Frame: Blood sample obtained at 26-30 weeks after a minimum of 7 injections and compliant with study protocol
Population: Subjects with available 26-30 week specimen (after 7 injections minimum) who were compliant with protocol up to the point of the blood draw. Included those with indicated preterm birth. . The subjects received either a 250 mg injection or a 500 mg injection and it is not relevant whether she was in the RCT or ancillary group. Those receiving the 250 mg dose include both the RCT and ancillary groups
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- 250 mg Dose: group received 250 mg dose
- 500 mg Dose: Group received 500 mg dose
Arm/Group | 250 mg Dose | 500 mg Dose
Number analyzed (Participants) | 66 | 55
ng/ml | 8.6 [6.8 to 11.5] | 16.2 [14.4 to 20.4]

7. Secondary Outcome: Preterm Birth by Dosing Group
Description: rate of preterm birth according to dosing group. Subjects were the same cohort in spec aims 1 and 2 . They were compliant with protocol, had a 26-30 week blood sample and did not miss more than 2 injections.
Time Frame: from enrollment till preterm delivery
Population: Those receiving the 250 mg dose include both the RCT and ancillary groups
Measure: Count of Participants; unit: Participants
Arm/Group | 250 mg Dose | 500 mg Dose
Number analyzed (Participants) | 54 | 62
Participants | 7 | 9

ADVERSE EVENTS:
Time Frame: Among those receiving either 250 mg or 500 mg OHPC adverse events were monitored from first injection until delivery for the mother up to 42 weeks gestation. This includes those with indicated preterm birth or absent blood sample but excluded those who were non-compliant, lost to followup, discontinued treatment or did not receive the drug.
Description: Adverse events are self reported by subjects and questioning was open ended without any direction by staff. Adverse events were analyzed by dose, the grouping by RCT or Ancillary is not relevant. Those receiving the 250 mg dose include both the RCT and ancillary groups. Subjects for this analysis included those with indicated preterm birth or absent blood sample but excluded those who were non-compliant, lost to followup, discontinued treatment or did not receive the drug.
Groups:
- 250 mg Dose: subject receiving 250mg of hydroxyprogesterone caproate
- 500 mg Dose: Pregnant subject receiving 500mg of hydroxyprogesterone caproate
- All Groups: all groups included Ancillary and both RCTs
Arm/Group | 250 mg Dose | 500 mg Dose | All Groups
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/66 | 0/131
Serious Adverse Events (participants affected / at risk) | 19/65 | 17/66 | 36/131
Other Adverse Events (participants affected / at risk) | 53/65 | 57/66 | 121/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 250 mg Dose (N=65) | 500 mg Dose (N=66) | All Groups (N=131)
suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) — Subject had suicidal ideation and was removed from study and drug stopped
SAEs unrelated to drug therapy (Pregnancy, puerperium and perinatal conditions) | 19 (19) | 16 (16) | 35 (35) — SAEs unrelated to drug therapy- these were related to hospital admission for pregnancy related issues
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 250 mg Dose (N=65) | 500 mg Dose (N=66) | All Groups (N=131)
injection site reaction (Musculoskeletal and connective tissue disorders) | 53 (53) | 57 (57) | 110 (110)
headache (Vascular disorders) | 24 (24) | 21 (21) | 43 (43)
nausea (Gastrointestinal disorders) | 17 (17) | 14 (14) | 31 (31)
diarrhea (Gastrointestinal disorders) | 12 (12) | 7 (7) | 19 (19)
vomiting (Gastrointestinal disorders) | 11 (11) | 4 (4) | 15 (15)
abdominal pain (Gastrointestinal disorders) | 10 (10) | 5 (5) | 15 (15)
constipation (Gastrointestinal disorders) | 7 (7) | 8 (8) | 15 (15)
dizziness (Nervous system disorders) | 7 (7) | 3 (3) | 10 (10)

LIMITATIONS AND CAVEATS:
Statistical analysis limited due to inadequate enrollment and subsequent small sample size and few cases of sPTB.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT03292731/Prot_SAP_019.pdf